CLINICAL TRIAL: NCT03060369
Title: BWH Critical Care Study of CareGuide for Evaluation of Emerging or Established Shock
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Reflectance Medical, Inc. (Unknown)
Responsible Party: Principal Investigator, Stephen D. Wiviott, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: BWH CareGuide
Record Dates: First submitted 2013-08-01; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Shock
Keywords: Tissue Perfusion; Noninvasive Monitoring; Near-infrared spectroscopy; CareGuide
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Established Shock (Cohort A): Meeting criteria i or ii, AND iii:
  i. SBP ≤ 90mm Hg for greater than 30 minutes ii. Requirement for vasopressor or ionotrope to maintain SBP > 90mm Hg iii. New dysfunction of at least one organ, including altered mental status, acute renal failure (increase from baseline in serum creatinine >0.3 mg/dL or by 50%), oliguria (<0.5 mL/kg/h for >6h) , or hepatic injury (ALT, AST, or total bilirubin >2xULN)suspected by the treating physician to be caused by organ hypoperfusion
  Interventions: Device: CareGuide™ device
- Emerging Shock (Cohort B): Meeting criteria i or ii, AND iii:
  i. New SBP ≤ 90mm Hg for greater than 30 minutes or recurrent shorter episodes, requiring use of or clinical anticipation of the need for fluid resuscitation or vasopressor/inotropic support to maintain SBP > 90 mm Hg ii. New dysfunction of at least one organ (as defined above), including altered mental status, acute renal failure, oliguria, or hepatic injury not explained by a specific non-hemodynamic cause iii. Does not meet criteria for Established Shock
  Interventions: Device: CareGuide™ device

INTERVENTIONS:
Device: CareGuide™ device — CareGuide™ is a minimal risk, non-invasive device that uses near-infrared spectroscopy to measure skeletal muscle oxygen saturation.

SUMMARY:
This pilot study aims to examine the relationship between continuously measured CareGuide™ muscle oxygen saturation (SmO2), tissue pH and data provided from standard monitoring techniques during the care of subjects with suspected established (Cohort A) or emerging (Cohort B) shock in the intensive care unit (ICU).

DETAILED DESCRIPTION:
Approximately 50 subjects meeting recruitment criteria will be enrolled with a minimum of 20 subjects meeting entry criteria for established shock (Cohort A).

Noninvasive near-infrared spectroscopy CareGuide™ measurements of SmO2, tissue pH and hematocrit will be collected from enrollment through device removal. These data will be compared to specific hemodynamic and laboratory parameters obtained as a part of routine care during the CareGuide™ monitoring period.

ELIGIBILITY:
Inclusion Criteria:

Subjects who are:

1. To be admitted to the intensive care unit
2. At least 18 years of age
3. Men or Women
4. Informed consent from subject or surrogate
5. Clinical diagnosis of established (Cohort A) or emerging (Cohort B) shock, as described above.

Exclusion Criteria:

Subjects with:

1. Body mass index >37
2. Trauma (primary diagnosis)
3. Pregnancy
4. Non-global conditions leading to regional increased lactate production (e.g. isolated thrombotic or embolic phenomena, limb, compartment syndrome)
5. Known untreated hypothyroidism
6. Known hypersensitivity to medical adhesives
7. Suspected carbon monoxide poisoning or methemoglobinemia
8. Goals of care restricting vital sign acquisition
9. Family member of investigators or study staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population is made up of adults admitted to an ICU with established or emerging shock.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Peak systemic lactate | Duration of monitoring (< 1 week)
  Cohort A

SECONDARY OUTCOMES:
Peak systemic lactate | Duration of monitoring (< 1 week)
  Cohort B
Temporal assessment of SmO2 and lactate | Duration of monitoring (< 1 week)
Standard hemodynamic measures stratified by shock type (cardiogenic, hypovolemic, distributive) | Duration of monitoring (< 1 week)
Systemic pH | Duration of monitoring (< 1 week)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided